CLINICAL TRIAL: NCT02555800
Title: Bevacizumab Versus Cidofovir for the Treatment of Recurrent Respiratory Papillomatosis: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Bevacizumab Versus Cidofovir for the Treatment of Recurrent Respiratory Papillomatosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro de Investigación en. Enfermedades Infecciosas, Mexico (Other Government)
Responsible Party: Principal Investigator, Gustavo Reyes-Teran, M.D., Centro de Investigación en. Enfermedades Infecciosas, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INER
Record Dates: First submitted 2015-08-12; First posted 2015-09-22 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Recurrent Respiratory Papillomatosis
Keywords: Laryngeal papillomatosis; Cidofovir; Bevacizumab; Recurrent respiratory papillomatosis
MeSH Terms: conditions — Recurrent respiratory papillomatosis; Laryngeal papillomatosis | interventions — Bevacizumab; Cidofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bevacizumab (Experimental): Patients will receive 3 intralesional injections of bevacizumab (Avastin, Genentech, San Francisco, California) every 3 to 6 weeks in a submucosal plane after surgical debulking. 12.5 mg of bevacizumab diluted in 3mL of 9% isotonic sodium chloride solution will be injected intralesionally using a 25 gauge.
  Interventions: Drug: Bevacizumab
- Cidofovir (Experimental): Patients will receive 3 intralesional injections of cidofovir every 3 to 6 weeks a submucosal plane after surgical debulking. 3.5 mL of cidofovir diluted to a concentration of 5 mg/mL in a 9% isotonic sodium chloride solution will be injected intralesionally using a 25 gauge.
  Interventions: Drug: Cidofovir
- Saline (Placebo Comparator): Patients will receive 3 intralesional injections of 3.5 mL of saline solution every 3 to 6 weeks in a submucosal plane after surgical debulking.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bevacizumab — Patients will receive 3 intralesional injections of bevacizumab (Avastin, Genentech, San Francisco, California) every 3 to 6 weeks in a submucosal plane after surgical debulking. 12.5 mg of bevacizumab diluted in 3mL of 9% isotonic sodium chloride solution will be injected intralesionally using a 25 gauge.
  Other Names: Avastin
  Arms: Bevacizumab
Drug: Cidofovir — Patients will receive 3 intralesional injections of cidofovir every 3 to 6 weeks a submucosal plane after surgical debulking. 3.5 mL of cidofovir diluted to a concentration of 5 mg/mL in a 9% isotonic sodium chloride solution will be injected intralesionally using a 25 gauge.
  Other Names: Vistide
  Arms: Cidofovir
Other: Placebo — Saline solution
  Arms: Saline

SUMMARY:
The aim of this study is to compare the efficacy of intralesional bevacizumab, a monoclonal antibody against vascular endothelial growth factor, versus the antiviral drug cidofovir in patients with recurrent respiratory papillomatosis.

DETAILED DESCRIPTION:
The investigators designed a randomized, double-blind, placebo-controlled study. Children and adults will be randomized to receive either 3 dosis of intralesional bevacizumab, cidofovir or saline solution. Primary endpoints are the assessment of changes in the annual surgery rate and Derkay papilloma severity grading scale; secondary endpoints are changes in the Voice Handicap Index and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with recurrent respiratory papillomatosis proven by biopsy.
* Patients with 2 or more previous surgeries for papillomatosis

Exclusion Criteria:

* Patients with heart or renal disease
* Patients who receive another adjuvant therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Changes in the annual surgery rate | 12 months
  Changes in the annual surgery rate before and after intervention
Severity of airway affection measured by the Derkay papilloma severity grading scale | 12 months
  Changes in the Derkay papilloma severity grading scale before and after intervention

SECONDARY OUTCOMES:
Hoarseness severity measured by the Voice Handicap Index | 12 months
  Changes in the Voice Handicap Index before and after intervention
Number of Treatment-Related Adverse Events According to Common Terminology Criteria for Adverse Events (CTCAE) | 12 months
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Reyes-Terán, M.D., Principal Investigator — Centro de Investigación en. Enfermedades Infecciosas, Mexico
Locations (1):
- Centro de Investigacion en Enfermedades Infecciosas, México, State of Mexico, Mexico

REFERENCES:
- [Derived] Ablanedo-Terrazas Y, Estrada-Camacho O, Alvarado-de la Barrera C, Ramirez-Garcia A, Tona-Acedo G, Bross-Soriano D, Schimelmitz-Idi J. Efficacy of cidofovir versus bevacizumab in recurrent respiratory papillomatosis: A randomized, double-blind, placebo-controlled pilot study. Acta Otorrinolaringol Esp (Engl Ed). 2022 Mar-Apr;73(2):82-88. doi: 10.1016/j.otoeng.2020.12.001. PMID 35397828